CLINICAL TRIAL: NCT03505333
Title: Liga Sure Versus Conventional Suture Ligature for Decrease Blood Loss During Abdominal Hysterectomy: Randomized Controlled Trial
Brief Title: Liga Sure Versus Conventional Suture Ligature for Decrease Blood Loss During Abdominal Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, lecturer, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: aswu/202/18
Record Dates: First submitted 2018-04-07; First posted 2018-04-23 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Decrease Blood Loss During Abdominal Hysterectomy

STUDY DESIGN:
Intervention Model Description: single-blinded randomized trials
Who Masked: Participant
Masking Description: Patients were randomized to two groups according to a two-blocked randomization list which was coded (a) or (b) at 1:1 ratio. The two parallel groups were prepared using a Computer-generated randomization system. The allocated groups were concealed in serially numbered sealed opaque envelopes that were opened only after recruitment. Patient allocation was performed prior to the induction of anesthesia by an independent researcher, who was not otherwise being involved in this study. The trial was appropriately single-blinded. The participants were blinded to the procedure performed.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional suture ligature (Experimental): use of conventional sutures for hysterectomy
  Interventions: Procedure: conventional suture
- Liga Sure (Active Comparator): use of conventional sutures plus use of Liga-sure for hysterectomy
  Interventions: Procedure: conventional suture

INTERVENTIONS:
Procedure: conventional suture — we use Liga-sure device for hysterectomy

SUMMARY:
Liga Sure represents a novel principle for hemostatic sealing of vessel-containing tissue based on feedback-programmed dosage of bipolar diathermy.(5) According to marketing of the device, Liga Sure has the potential to replace the use of conventional suture ligature within a broad range of surgical procedures, also including removal of the uterus. While the use of Liga Sure has been critically assessed for a range of procedures such as hemorrhoidectomy, splenectomy, bile duct, urological and gastric operations,(6-12) a similar scientific evaluation of its suitability for abdominal removal of the uterus is lacking in the literature. The most promising aspect of Liga Sure in hysterectomy is the potential shorter operation time and decrease blood loss. Because removal of the uterus traditionally is the most frequently performed major gynecological operation,(13) the introduction of a time-sparing new technique could have significant impact on resource consumption.

The aim of the study:

we aimed at evaluating the use of Liga Sure compared with conventional suture ligature during abdominal hysterectomy, in a prospective randomized controlled trial with special emphasis on the safety, the duration of the procedure and the amount of blood loss.

DETAILED DESCRIPTION:
Hysterectomy represents the second most performed surgery in gynecology after the Cesarean Section. Worldwide most of the hysterectomies are performed abdominally. (1) One in 9 women will undergo a hysterectomy in their lifetime. (1) Surgical blood loss of more than 1000 mL or blood loss that requires a blood transfusion usually defines intraoperative hemorrhage. Intraoperative hemorrhage has been reported in 1% to 2% of hysterectomy studies. (2) As with any surgical treatment, complications affect the outcomes of hysterectomy. Hemorrhage, which is the most frequent and critical complication, often occurs during surgery. Data from The Danish Hysterectomy and Hysteroscopy Database (DHHD) has revealed a relatively high complication rate of 16-18% from 1998 to 2006, of which perioperative bleeding complications represent the most common cause.(3 )From 2004 to 2006, 6-8% of all women undergoing benign hysterectomy in Denmark experienced a bleeding complication .(4 ) Therefore, adequate hemostatic techniques are essential during abdominal hysterectomy. Currently, surgical hemostasis can be secured by a variety of methods, including mechanical sutures (or clamping), electric coagulation, ultrasonically activated scalpel or drugs. (4)

Liga Sure represents a novel principle for hemostatic sealing of vessel-containing tissue based on feedback-programmed dosage of bipolar diathermy.(5) According to marketing of the device, Liga Sure has the potential to replace the use of conventional suture ligature within a broad range of surgical procedures, also including removal of the uterus. While the use of Liga Sure has been critically assessed for a range of procedures such as hemorrhoidectomy, splenectomy, bile duct, urological and gastric operations,(6-12) a similar scientific evaluation of its suitability for abdominal removal of the uterus is lacking in the literature. The most promising aspect of Liga Sure in hysterectomy is the potential shorter operation time and decrease blood loss. Because removal of the uterus traditionally is the most frequently performed major gynecological operation,(13) the introduction of a time-sparing new technique could have significant impact on resource consumption.

The aim of the study:

we aimed at evaluating the use of Liga Sure compared with conventional suture ligature during abdominal hysterectomy, in a prospective randomized controlled trial with special emphasis on the safety, the duration of the procedure and the amount of blood loss.

Materials and Methods After obtaining ethics committee approval and patient consent, we will randomize patients about to undergo elective abdominal hysterectomy, between the use of Liga Sure and conventional suture ligature during the operation. Patients who were admitted for non-acute planned abdominal total or subtotal hysterectomy were eligible. Two experienced lecturer gynecologists performed the operations. 60 patients for each of the tow operators were block-randomized. The treatment options, 30 of each in each randomization block, were first concealed in envelopes. Thereafter, the sequence was generated using computer-generated random number lists. The 60 projected patients will include and will be randomized between December 2017 and December 2019. The following pre- and intra-operative parameters will be registered: the indication for the operation, the type of incision, procedures in addition to the hysterectomy, the duration of the operation, the blood loss and the use of intra-operative blood transfusions. When Liga Sure was used, the eventual number of its replacements by suture ligature due to unsuccessful vessel sealing was registered. During the first 30 post-operative days, the following parameters were registered: all types of re-operations, the use of blood transfusion, the occurrence of fever above 38°C, all types of infections, deep vein thrombosis and the length of the post-operative hospital stay.

Measurement of Blood Loss Blood loss well be estimated by a combination of direct measurement and gravimetric method (14). The direct measurement well performed by collecting most of the lost blood into a suction bottle using a suction apparatus. Care was taken to collect most of (if not all) the amniotic fluid in a separate suction bottle. The gravimetric method well used to estimate the amount of blood loss in the surgical towels. The dry surgical towels (40 by 40 cm) were weighed before surgery. Intraoperatively, the towels were used to dry up all the blood in the surgical field then these towels were collected into a sterile metallic bowl which was weighed empty before surgery. When 5 soaked towels are collected in the bowl, the bowl with the collected soaked towels are handled to the circulating nurse to weigh it by a highly accurate digital balance and then calculate the amount of blood loss in the towels by the following formula: amount of blood loss in the soaked towels (in ml) = weight of the metallic bowl with the collected soaked towels in it (in gm)- [weight of the empty bowel (in gm) + weight of the towels before surgery (in gm)]. The collected blood in the suction bottle well added to the total calculated amount of blood loss in the towels.

The primary outcomes are the total blood loss during and after hysterectomy. the secondary outcome is another surgical maneuver to decrease blood loss (need of suturing in the Liga sur arm), operative time ,any complication Statistical Analysis; Continuous variables were presented as mean ± standard deviation, while categorical variables were presented as frequencies and percentages. The IBM (SPSS) Statistics, version 20.0, for Windows was used for statistical analysis. P values ≤0.05 were considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* patient prepared for an elective benign hysterectomy

Exclusion Criteria:

1. Patients with a cardiac, hepatic, renal or thromboembolic disease.
2. patients with pelvic endometriosis and adnexal mass.
3. patients with endometrial or cervical cancer
4. radical hysterectomy

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 90 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
decrease blood loss during hysterectomy | intra-operative
  Blood loss well be estimated by a combination of direct measurement and gravimetric method

SECONDARY OUTCOMES:
need for blood transfusion, | intraoperative
  number RBC unit trasfused
post operative HB | 24 hour post operative
  measure HB pos operative
operative time | intra operative
  time of operation

CONTACTS AND LOCATIONS:
Overall Officials: hany f sallam, md, Principal Investigator — Aswan University Hospital
Locations (1):
- AswanUH, Aswān, Egypt